CLINICAL TRIAL: NCT04638582
Title: Phase II Randomized Controlled Trial of Neoadjuvant Pembrolizumab or Pembrolizumab With Histology-Specific Chemotherapy for Operable Stage IA3 to IIA Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pembrolizumab as Neoadjuvant Therapy for Resectable Stage IA3 to IIA Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jonathan Spicer, Assistant Professor of Surgery, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK3475-A74
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: Non-Small Cell Lung Cancer; Immunotherapy; Immune Checkpoint Inhibition; Early Stage Lung Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant pembrolizumab + adjuvant pembrolizumab +/- adjuvant chemotherapy (Experimental): Neoadjuvant: Participants receive pembrolizumab [200 mg, intravenous (IV)] every 3 weeks for 3 cycles.
  Adjuvant: Participants receive pembrolizumab [400 mg IV] every 6 weeks for 6 cycles, and may receive histology-specific adjuvant chemotherapy [consisting of carboplatin AUC 6 and paclitaxel 200 mg/m2, or carboplatin AUC 5 and paclitaxel 500 mg/m2] every 3 weeks for 4 cycles, if indicated.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed
- Neoadjuvant pembrolizumab and chemotherapy + adjuvant pembrolizumab +/- adjuvant chemotherapy (Experimental): Neoadjuvant: Participants receive pembrolizumab [200 mg, intravenous (IV)] every 3 weeks for 3 cycles in combination with standard of care histology-specific chemotherapy [consisting of carboplatin AUC 6 and paclitaxel 200 mg/m2, or carboplatin AUC 5 and paclitaxel 500 mg/m2] every 3 weeks for 3 cycles.
  Adjuvant: Participants receive pembrolizumab [400 mg IV] every 6 weeks for 6 cycles, and may receive histology-specific adjuvant chemotherapy [consisting of carboplatin AUC 6 and paclitaxel 200 mg/m2, or carboplatin AUC 5 and paclitaxel 500 mg/m2] every 3 weeks for 4 cycles, if indicated.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — Neoadjuvant pembrolizumab 200 mg IV every 3 weeks, given on cycle day 1. Adjuvant pembrolizumab 400 mg IV every 6 weeks, given on cycle day 1.
  Other Names: Keytruda; MK-3475
Drug: Carboplatin — Carboplatin AUC 6 IV (maximum dose: 900 mg) for squamous cell carcinoma, and AUC 5 IV (maximum dose: 750 mg) for non-squamous cell carcinoma, every 3 weeks, given on cycle day 1.
Drug: Paclitaxel — Paclitaxel 200 mg/m2 IV every 3 weeks, given on cycle day 1. Only given to participants with squamous cell carcinoma.
Drug: Pemetrexed — Pemetrexed 500 mg/m2 every 3 weeks, given on cycle day 1. Only given to participants with non-squamous cell carcinoma.

SUMMARY:
This is a prospective, randomized, single-site, open-label Phase II trial of neoadjuvant pembrolizumab (3 cycles) followed by surgery, versus concomitant neoadjuvant pembrolizumab with platinum doublet chemotherapy (3 cycles) followed by surgery for participants with Stage IA3, IB and IIA non-small-cell lung cancer (NSCLC). Participants will be offered pembrolizumab (6 cycles), and standard of care adjuvant chemotherapy (4 cycles) if applicable.

DETAILED DESCRIPTION:
The use of ctDNA levels and resolution in relation to treatment response has been studied in various types of cancer, notably melanoma, colorectal and pancreatic cancers. In pancreatic cancer, it was particularly noted to be useful for the prediction of recurrence and survival patterns. In NSCLC, there is a growing need to identify patients who are more likely to respond to immunotherapies given the rates of recurrence, and ctDNA was described to be a useful tool in the prediction of pathological response in this population. In fact, ctDNA was shown to correlate with disease resolution in NSCLC and higher levels of ctDNA in non-responding patients.

The central research question of this trial is focused on the ability to predict the occurrence of a pCR based on resolution of ctDNA detectability in early stage NSCLC. The biomarker collection plan will provide tumor and plasma samples from which whole exome sequencing will be performed to monitor disease response. The endpoint is focused on the elimination of ctDNA (both replicates = 0%) at the completion of systemic therapy, prior to surgical resection. All patients will be re-tested for ctDNA levels 30 days post-surgery to determine if those patients who did not experience ctDNA resolution after systemic therapy will experience resolution with the addition of surgery.

With the ctDNA treatment response arc, the investigators will be able to address the primary objective of the study: to establish ctDNA levels in early stage NSCLC as a reliable measure of local disease burden in the context of systemic therapy, with the lower end of the detection limit correlating to the extent of pathological response. The investigators hypothesize that in a cohort of patients with stage IA3, IB and IIA NSCLC, pre-operative pembrolizumab with or without histology-specific chemotherapy will cause resolution of ctDNA detectability that correlates with a pathological complete response (pCR) to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed (by core biopsy) NSCLC and histologically confirmed stages IA3, IB and IIA NSCLC (AJCC 8th edition).
* Able to undergo protocol therapy, including necessary surgery.
* If female: may participate if no active pregnancy, not breastfeeding, and at least one of the following: is not a woman of childbearing potential (WOCBP), or is a WOCBP using contraceptive methods.
* If male: must agree to refrain from donating sperm, and must either be abstinent or agree to use contraception.
* ECOG 0-1
* Available formalin-fixed paraffin embedded (FFPE) tumor tissue samples

Exclusion Criteria:

* Has one of the following tumor locations/types: NSCLC involving the superior sulcus, large cell neuroendocrine cancer (LCNEC) or sarcomatoid tumor.
* History of immunodeficiency, HBV, HCV, HIV. No HBV, HCV or HIV testing is required unless mandated by local health authority.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has had an allogenic tissue/solid organ transplant.
* Has a known severe hypersensitivity (≥ Grade 3) to pembrolizumab, its active substance and/or any of its excipients. (Refer to the respective Investigator's Brochure for a list of excipients.)
* Has a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents and/or to any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
* Has received colony-stimulating factors (eg, G-CSF, GM-CSF or recombinant erythropoietin) within 2 weeks before randomization
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anticancer therapy including investigational agents for the current malignancy prior to randomization/allocation.
* Has received prior radiotherapy within 2 weeks of start of trial treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of trial drug. Note: killed vaccines are allowed.
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (dose exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial drug.
* Has a known additional malignancy that is progressing or requires active treatment within the past (5 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-08-28 (Actual); Primary Completion 2025-08-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
ctDNA resolution | Up to 2 years
  ctDNA resolution is defined as the change or resolution in tumor-derived DNA found in the bloodstream from diagnosis to after neoadjuvant therapy and after surgery, correlated with pathological complete response (pCR).

SECONDARY OUTCOMES:
Imaging measures of response | Up to 3 years
  Imaging measures of response is defined as individual measures of response for conventional CT (quantification of response by RECIST 1.1 criteria), PET (change in standardized uptake values [SUV]) and diffusion-weighted MRI (change in apparent diffusion coefficient [ADC] obtained by image analysis software package), in correlation with pathological complete response (pCR).
Pathological complete response (pCR) rate | Up to 3 years
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
Major pathological response (MPR) rate | Up to 3 years
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.
Adverse event (AE) rate | Up to 3 years
  Number of participants experiencing AEs will be recorded. An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Perioperative complications rate | Up to 3 years
  Number of participants experiencing perioperative complications will be recorded.

OTHER OUTCOMES:
Overall survival (OS) | Up to 3 years
  OS is defined as the time from randomization to death due to any cause.
Disease-free survival (DFS) | Up to 3 years
  DFS is defined as the time from initial treatment to the first of the following events: disease or local progression, inability to resect tumor, local or distant recurrence, or death.
Anatomical segmentectomy rate | Up to 3 years
  Number of participants undergoing an anatomical segmentectomy will be recorded. An anatomical segmentectomy is defined as surgery based on the lung segments, 10 on the right lung, 8 on the left lung, with each segment having different morphology, size and blood vessel branch.
Single cell RNA sequencing (scRNAseq) | Up to 3 years
  scRNAseq is defined as complete transcriptomic data from tumor epithelial, stromal and immune compartments obtained from tumor samples.
Imaging mass cytometry (IMC) panel analyses | Up to 3 years
  IMC panel is performed on tumor core biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Spicer, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No